CLINICAL TRIAL: NCT04064593
Title: SDB Prevalence and Cardiovascular Outcomes of MI Survivors
Brief Title: Sleep Disordered Breathing (SDB) Prevalence and Cardiovascular Outcomes of Myocardial Infarction (MI) Survivors
Acronym: AMISLEEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P171101J
Record Dates: First submitted 2019-08-05; First posted 2019-08-22 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Acute Myocardial Infarction; Sleep Apnea
Keywords: Acute Myocardial Infarction; Sleep Apnea; Outcomes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polygraphy (Experimental)
  Interventions: Diagnostic Test: Polygraphy

INTERVENTIONS:
Diagnostic Test: Polygraphy — The polygraphy consists of recording during sleep, respiratory flow by mean of a nasal cannula, respiratory movement by mean of a thoracic belt with inductance plethysmography, blood oxygenation and heartbeats by a fingertip transcutaneous oxymetry.
  Starting and ending of the recording will be programmed based on patient interview regarding usual sleep hours.
  Polygraphy data are anonymized before being sent to the Cloud and therefore to the core lab.
  Polygraphic data will be scored in centralized manner.
  Results of the polygraphy will be sent to the cardiology department with advice for treatment and follow-up.
  If necessary, the core-lab will provide tele-counseling regarding SDB management.

SUMMARY:
The AMISLEEP study is nested in the "FRENCHIE" registry.

The objective is to use routine clinical and polygraphic data to capture SDB/SAS (Sleep Disordered Breathing/Sleep Apnea Syndrome) physiological heterogeneity in relation to clinically relevant cardiovascular outcomes.

Specifically, the investigators hypothesize that unique clusters (phenotypes) of patients could be identified by applying unsupervised learning methods to these data and that the clusters would be differentially associated with risk of adverse cardiovascular outcomes (ACS), TIA, stroke or death). The ultimate goal is to identify patients more at risk that could be included in interventional studies that would test whether SDB/SAS treatment can improve this risk.

DETAILED DESCRIPTION:
All patients included in the "FRENCHIE" registry (Acute Myocardial Infarction (AMI) patients hospitalized within 48h from symptom onset) are eligible, and will be asked for their written informed consent for this nested study in case of the absence of any non-inclusion criteria.

Baseline clinical examination and laboratory tests are based on the usual care and are those collected in "FRENCHIE".

A simplified polygraphy is performed during the hospitalization for AMI. Starting and ending of the recording will be programmed based on patient interview regarding usual sleep hours.

Together with the polygraphy, questionnaires will be given to the patient regarding general sleep quality

Polygraphic data will be scored in centralized manner. Results of the polygraphy will be sent to the cardiology department with advice for treatment and follow-up. If necessary, the core-lab will provide tele-counseling regarding SDB management to centers.

Follow-up will be performed through the national administrative databases, as in the "FRENCHIE" registry.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in FRENCHIE registry (cf. NCT04050956 for FRENCHIE registry's selection criteria)
* Signed consent for AMI-Sleep study

Exclusion Criteria:

* Patient under treatment for SDB/SAS prior to its inclusion in FRENCHIE registry
* Cognitive disorientation and communicative disabilities (left to investigator's discretion) not able to fill-out a questionnaire
* Severe diseases with anticipated mortality less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2007 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Contribution of SDB/SAS to events after AMI | 12 months follow up
  Contribution of SDB/SAS to incident cardiovascular events and mortality during the first year following acute myocardial infraction :
  Cardiovascular event will be defined as incident acute coronary syndrome (ACS), transient ischemic attack (TIA), stroke or death of any cause after discharge during the first year following the AMI event. Time from discharge to the first event will be considered.

SECONDARY OUTCOMES:
Associations between presence, type and severity of SDB and the severity of the initial coronary disease | Through the end of hospitalization, an average of 5 days
  The severity of the index event (number of stents combined with revascularizations and coronary bypass) will be compared to type and severity of SDB (apnea-hypopnea index AHI), to evaluate if both are associated
Validate the Berlin questionnaire to screen for obstructive and central SDB/SAS in the AMI patients | Through the end of hospitalization, an average of 5 days
  Concordance between the result of the Berlin questionnaire and the presence of obstructive SDB/SAS measured by polygraphy as reference and concordance between the result of the Berlin questionnaire and the presence of central SDB/SAS measured by polygraphy as reference.
Evaluate health care related costs during the year following hospital discharge. | 12 months follow up
  Health care related costs for SDB considered will be: confirmation of SDB by an additional polysomnography, SDB treatments.
Comparison of health care consumption between SDB and non-SDB patients | 12 months follow up
  Health care consumption and health care related costs will be compared between patients :
  * without SDB
  * with mild SDB (AHI between 5 and 14/h)
  * with moderate SDB (AHI between 15h to 29/h)
  * with severe SDB (AHI ≥ 30/h)
  Health care consumption and health care related costs considered will be AMI recurrence, incident TIA/stroke, cardiac arrhythmia, heart decompensation, diabetes, depression and cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Gabriel STEG, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Duran J, Esnaola S, Rubio R, Iztueta A. Obstructive sleep apnea-hypopnea and related clinical features in a population-based sample of subjects aged 30 to 70 yr. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):685-9. doi: 10.1164/ajrccm.163.3.2005065. PMID 11254524
- [Background] Crawford-Achour E, Dauphinot V, Martin MS, Tardy M, Gonthier R, Barthelemy JC, Roche F. Protective Effect of Long-Term CPAP Therapy on Cognitive Performance in Elderly Patients with Severe OSA: The PROOF Study. J Clin Sleep Med. 2015 Apr 15;11(5):519-24. doi: 10.5664/jcsm.4694. PMID 25700873
- [Background] Cadelis G, Fayad Y Monteagudo OE. [Prevalence of symptoms and risk of obstructive sleep apnea syndrome assessed by the Berlin Questionnaire among professionals of a health facility]. Rev Epidemiol Sante Publique. 2016 Dec;64(6):405-414. doi: 10.1016/j.respe.2016.06.332. Epub 2016 Oct 31. French. PMID 27810127
- [Background] Tishler PV, Larkin EK, Schluchter MD, Redline S. Incidence of sleep-disordered breathing in an urban adult population: the relative importance of risk factors in the development of sleep-disordered breathing. JAMA. 2003 May 7;289(17):2230-7. doi: 10.1001/jama.289.17.2230. PMID 12734134
- [Background] Heinzer R, Vat S, Marques-Vidal P, Marti-Soler H, Andries D, Tobback N, Mooser V, Preisig M, Malhotra A, Waeber G, Vollenweider P, Tafti M, Haba-Rubio J. Prevalence of sleep-disordered breathing in the general population: the HypnoLaus study. Lancet Respir Med. 2015 Apr;3(4):310-8. doi: 10.1016/S2213-2600(15)00043-0. Epub 2015 Feb 12. PMID 25682233
- [Background] Levendowski D, Steward D, Woodson BT, Olmstead R, Popovic D, Westbrook P. The impact of obstructive sleep apnea variability measured in-lab versus in-home on sample size calculations. Int Arch Med. 2009 Jan 2;2(1):2. doi: 10.1186/1755-7682-2-2. PMID 19121211
- [Background] Jesus EV, Dias-Filho EB, Mota Bde M, Souza Ld, Marques-Santos C, Rocha JB, Oliveira JL, Sousa AC, Barreto-Filho JA. Suspicion of obstructive sleep apnea by Berlin Questionnaire predicts events in patients with acute coronary syndrome. Arq Bras Cardiol. 2010 Sep;95(3):313-20. doi: 10.1590/s0066-782x2010005000103. Epub 2010 Aug 6. PMID 20676583
- [Background] Gus M, Goncalves SC, Martinez D, de Abreu Silva EO, Moreira LB, Fuchs SC, Fuchs FD. Risk for Obstructive Sleep Apnea by Berlin Questionnaire, but not daytime sleepiness, is associated with resistant hypertension: a case-control study. Am J Hypertens. 2008 Jul;21(7):832-5. doi: 10.1038/ajh.2008.184. Epub 2008 May 1. PMID 18451807
- [Derived] Balagny P, D'Ortho MP, Berard L, Rousseau A, Gourmelen J, Ravaud P, Durand-Zaleski I, Simon T, Steg PG; AMI SLEEP investigators. AMI-Sleep: protocol for a prospective study of sleep-disordered breathing/sleep apnoea syndrome and incident cardiovascular events after acute myocardial infarction. BMJ Open. 2025 Feb 18;15(2):e090093. doi: 10.1136/bmjopen-2024-090093. PMID 39965954